CLINICAL TRIAL: NCT04487353
Title: Development And Use Of Virtual Reality Application In Teaching Birth Mechanism
Brief Title: Teaching the Mechanism of Birth by Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Karabuk University (Other)
Responsible Party: Principal Investigator, Sebahat Hüseyinoğlu, Prelector (principal investigator), Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020/256
Record Dates: First submitted 2020-07-11; First posted 2020-07-27 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Educational Problems
Keywords: virtual reality

STUDY DESIGN:
Intervention Model Description: The sample will consist of 105 midwifery students, 35 control, 35 experiment I and 35 experiment II, as a result of the G-power analysis calculated from 0.95 power, among the midwifery students who took the birth mechanism 4 hours theoretically in their curriculum within the scope of normal birth lesson.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment Group (Experimental): The Labor Evaluation Information Scale (LEIS) was administered as a pre-test before applying to 30 students who had taken a course on childbirth. After the pre-test, the application was carried out with the "Labor mechanism application developed with virtual reality technology (VRT-LMA)". Immediately after the application, data were collected with the "LEIS", "sense of presence scale" and "cognitive load scale". Post-test was performed again with the Labor Evaluation Information Scale (LEIS) 5 weeks after the application.
  Interventions: Other: Labor mechanism application developed with virtual reality technology (VRT-LMA)
- Control Group (No Intervention): Before the theory training, the Assessment Knowledge Scale (LEIS) was administered as a pre-test to 31 students in the control group who had taken a course on obstetrics. After the pre-test, theory training including birth knowledge was given. "Labor mechanism application developed with virtual reality technology (VRT-LMA)" was not applied to the control group. After 4 hours of theoretical training, the final test was performed using LEIS. After 5 weeks, the last test was repeated.

INTERVENTIONS:
Other: Labor mechanism application developed with virtual reality technology (VRT-LMA) — In phase I: VRT-LMA application was developed. (Female in lithotomy position, bony pelvis, flexion of the coccyx back about 2 cm and the Hodge plane were modeled as lines. The theory training to be given to the control group was prepared in accordance with the curriculum.
  II. In the first stage: Pre-test was applied to both groups. After the pretest, theory training was given to the control group and the posttest was applied. VRT-LMA was applied to the experimental group, and the posttest, sense of presence scale, and cognitive load scale were administered.
  II. In the first stage: Pre-test was applied to both groups. After the pretest, theory training was given to the control group and the posttest was applied. VRT-LMA was applied to the experimental group, and the posttest, sense of presence scale, and cognitive load scale were administered.
  III. In the second stage: the post-test and analyzes were performed after 5 weeks in both groups.
  Arms: Experiment Group

SUMMARY:
With the virtual birth application,

* Learning the physiology and mechanism of birth,
* To monitor the progress of birth and to understand deviations from normal,
* Learning normal birth,
* It will provide the opportunity to see all the emergencies that may be encountered at birth and besides these, the information will be remembered for a long time.

In this way, the effectiveness of virtual birth in midwifery education will be evaluated.

Teaching the birth, which is one of the cornerstones of midwifery education and where the students find the opportunity to practice clinically, with virtual reality application, will minimize clinical application errors and will provide early diagnosis of adverse conditions such as fetal presentation and placental anomalies that may occur at birth. It is an up-to-date and important subject that will enable them to see the stages of birth in three dimensions with the virtual delivery application without any obstacle in midwifery education, the birth process, the birth mechanisms of the baby from the birth canal.

DETAILED DESCRIPTION:
In recent years, many studies have shown that technology assisted learning is a new learning approach (1); In particular, learning environments involving virtual reality (VR) techniques have become a powerful tool for educators and students (3, 4). Significant progress has been made in various fields, enabling students to interact with the virtual world. These technologies support many educational activities originally offered in web-based learning environments. In midwifery education, the use of simulation has become an important training method in the last decade (2). Simulation is a method that reflects a clinical situation as close to reality as possible, making it easier to understand and manage when this situation is actually encountered in clinical practice. Ensuring patient safety, efforts to increase students' competence have enabled the use of simulation to become more widespread in the training of health professionals (5). Using virtual reality in midwifery education will enable students to use midwifery practices effectively before going to clinical practice. Teaching the birth, which is one of the cornerstones of midwifery education and where the students find the opportunity to practice clinically, with virtual reality application, will minimize clinical application errors and will provide early diagnosis of adverse conditions such as fetal presentation and placental anomalies that may occur at birth.

Type of the Study: The study is an experimental study planned as an experimental and control group.

The research consists of 2 parts. In Part I, Virtual Reality Application will be Developed. Virtual birth software will be prepared through service procurement. For this, algorithms will be created by the researchers by writing in detail the physiology, stages, mechanism and anatomy of the woman in detail.

II. The application of the research will be done in the department.

SECTION I: Development of Virtual Reality Application

In the 1st part of the research, virtual birth software will be prepared through service procurement. For this, algorithms will be created by the researchers by writing in detail the physiology, stages, mechanism and anatomy of the woman in detail. This algorithm will be transferred to the glasses based on the images and drawings of the anatomy of the woman from the birth atlases and the real images shared on the internet at the moment of birth. As stated in the budget form, services will be procured for the development of the virtual birth software.

With the virtual birth application,

* To learn the physiology and mechanism of birth,
* To monitor the progress of the birth and to understand deviations from the normal,
* Learning normal birth,
* It will provide the opportunity to see all the emergencies that may be encountered at birth and besides these, the information will be remembered for a long time. In this way, the effectiveness of virtual birth in midwifery education will be evaluated.

II. Department: Application of the Research

In this last part of the research, the application part of the research has been started. The research will consist of 3 groups, 2 experimental groups and a control group. 35 students will be admitted to each group as a result of G-power analysis calculated with 0.95 power.

The Universe of the research will consist of 464 Midwifery students studying at Karabük University.

The sample will consist of 105 midwifery students, 35 control, 35 experiment I and 35 experiment II, as a result of the G-power analysis calculated by 0.95 power, among midwifery students who took the birth mechanism 4 hours theoretically in their curriculum within the scope of normal birth lesson.

At the first stage: after 4 hours of theory training for all three groups, the information form (DEDBF) to be prepared by the researchers to be used in this research will be applied as the first test.

In the second stage: No application will be made to the control group, computer-aided and guided virtual reality application will be applied to the experimental group, and computer-free and non-guided virtual application will be monitored to the experimental group II.

In the third stage: DEDBF questions will be replaced and posttests will be applied. After the 4-hour theory training for the control group, the post-test will be done after the virtual birth application is watched on the experiment groups. Also, at this stage, "Cognitive Load Scale" and "Feel of Inventory" will be applied to the experimental groups after the application.

In the fourth stage: After three weeks, the DEDBF will be applied again to the three groups, and the effectiveness of the application of virtual birth will be examined in recalling and recalling the information.

During applications, experiment and control group videos and images will be taken and published visually in the thesis.

Students who could not participate in the study and were selected as a control group in randomization will also be provided with virtual reality glasses after the study, so that all students will see the virtual birth application and equality will be achieved.

Data Collection Tools:

Data collection form: It is planned to apply a form consisting of 15 questions, which includes the characteristics of the participants such as age, marital status, educational status and family type.

Birth Action Assessment Information Scale (DEDBF): The scale will be prepared by the researchers themselves for use in this thesis. For the preparation of the form, the latest literature information was reviewed by the researchers, the midwifery core curriculum (EUÇEP) created by YÖK, and a 42-question information form containing items on the physiology, stages and mechanism of delivery was prepared. The items in the information form will be presented to the students in the form of a full sentence that can be true or false, and students will be asked to answer these statements as "True" or "False". Total response time is 30 minutes. Correct answers will be evaluated as 1 point, Wrong answers will be evaluated as 0 points. Wrong expressions were also used in the information form, and these items were coded in reverse compared to others. The lowest score to be taken from the information form is 0 and the highest total score is 42.

Cognitive Load Scale: Kılıç et al. (2004) "Cognitive Load Scale" (BYÖ) adapted to Turkish will be used. It has single factor and nine points (very little, very little, little, partly little, neither more nor less, more, more, more, more, more, more or more). The Cronbach Alpha internal consistency coefficient of the original version was found to be .90 (7). Kılıç et al. (2004) in the adaptation study, the Cronbach Alpha internal consistency coefficient was found as .78. The lowest point of the scores obtained from the scale is 1.00, the middle point is 5.00 and the highest point is 9.00. Participants scoring less than five points were evaluated as "cognitively overloaded", and participants scoring higher than five points were evaluated as "cognitively overloaded".

Availability Sensitivity Scale: It is the scale whose original validity in Turkish was valid in 2018 by Gökoğlu et al. The scale is measured in virtual reality based learning environments. The scale has 5 factors (subscale), namely Participation (Factor 1), Cohesion / Surrounding (Factor 2), Sensory Commitment (Factor 3), Interaction (Factor 4) and Interface Quality (Factor 5) and consists of 29 questions (8 ). According to the exploratory factor analysis (AFA) and confirmatory factor analysis (CFA), the total variance explained by the 5-factor structure was 41.197% and the reliability coefficient of the scale was .844.

Data Analysis of the Research: Analysis of the data of the study will be done using IBM SPSS for Mac book 24 version.

ELIGIBILITY:
Inclusion criteria for the study; Being a 4th year student of Health Sciences University, Gulhane Health Sciences Faculty, Midwifery Department, Volunteering to participate in research Exclusion criteria from the study; Being a first year student. being a second year student being a third year student

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Labor Evaluation Information Scale (LEIS) | within 6 weeks
  To measure the knowledge level of both groups about the mechanism of labor. To compare the changes in the knowledge level of students who have experienced VRT-LMA and students who have only theory education.

SECONDARY OUTCOMES:
Cognitive Load Scale | within 6 weeks
  At this stage, "Cognitive Load Scale" will be applied to the experimental groups after the application.
  It has single factor and nine points (very little, very little, little, partially little, neither more nor less, more, more, more, more, more, more). The Cronbach Alpha internal consistency coefficient of the original version was found to be .90 (7). Kılıç et al. (2004) in the adaptation study, the Cronbach Alpha internal consistency coefficient was found as .78. The lowest point of the scores obtained from the scale is 1.00, the middle point is 5.00 and the highest point is 9.00. Participants who scored below five points were evaluated as "cognitively overloaded", and participants who scored above five points were evaluated as "cognitively overloaded".
Availability Sensitivity Scale | within 6 weeks
  At this stage, "Availability Sensitivity Scale" will be applied to the experimental groups after the application. Availability Sensitivity Scale: It is the scale whose original validity in Turkish was valid in 2018 by Gökoğlu et al. The scale is measured in virtual reality based learning environments. The scale has 5 factors (subscale), namely Participation (Factor 1), Cohesion / Surrounding (Factor 2), Sensory Commitment (Factor 3), Interaction (Factor 4) and Interface Quality (Factor 5) and consists of 29 questions (8 ). According to the exploratory factor analysis (AFA) and confirmatory factor analysis (CFA), the total variance explained by the 5-factor structure was 41.197% and the reliability coefficient of the scale was .844. It is scored from 1 to 5. 1 ever, 5 are listed as completely.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'm undecided now. I want to decide in the future

REFERENCES:
- [Background] Cooper S, Cant R, Porter J, Bogossian F, McKenna L, Brady S, Fox-Young S. Simulation based learning in midwifery education: a systematic review. Women Birth. 2012 Jun;25(2):64-78. doi: 10.1016/j.wombi.2011.03.004. Epub 2011 Apr 13. PMID 21489894
- [Background] Bjerrum AS, Hilberg O, van Gog T, Charles P, Eika B. Effects of modelling examples in complex procedural skills training: a randomised study. Med Educ. 2013 Sep;47(9):888-98. doi: 10.1111/medu.12199. PMID 23931538
- See also: Şendir, M. (2013). Kadın Sağlığı Hemşireliği Eğitiminde Simülasyon Kullanımı. F.N. Hem. Dergisi, 21 (3), 205-212. — https://www.researchgate.net/profile/Merdiye_Sendir/publication/260591472_Kadin_Sagligi_Hemsireligi_Egitiminde_Simulasyon_Kullanimi-_Use_of_Simulation_in_Women's_Health_Nursing_Education/links/0f317531a20c09f9fa000000/Kadin-Sagligi-Hemsireligi-Egitiminde-Simulasyon-Kullanimi-Use-of-Simulation-in-Womens-Health-Nursing-Education.pdf
- See also: Kılıç, A. G. E., & Karadeniz, Ö. G. Ş. (2004). Hiper ortamlarda öğrencilerin bilişsel yüklenme ve kaybolma düzeylerinin belirlenmesi. Kuram ve Uygulamada Eğitim Yönetimi, 40(40), 562-579. — https://dergipark.org.tr/en/pub/kuey/issue/10357/126808